CLINICAL TRIAL: NCT04431700
Title: Impact of Anti-Inflammatory Whole-Food Diet in Crohn's Disease and Predicting Response to Therapy
Brief Title: Study of Dietary Composition in Crohn's Disease
Acronym: CD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete enrollment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001120
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
Keywords: Crohn's Disease; IBD; Anti-inflammatory Diet
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Diet

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, controlled trial. All eligible participants will be randomly assigned to one of two diets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory whole food (Experimental): Included food items will include a defined minimum diversity of fruits, vegetables, and nuts based on complementary phytonutrient contents, particularly those rich in phenolic compounds such as ellagitannins and sulforaphanes. Selected herbs (e.g., curcumin), fermented foods, fats (e.g., avocado), and oils (e.g., olive oil) will be permitted or encouraged. Recommended portions of complex carbohydrates (50% - 60%) and lean proteins (20% - 30%) will form the basis of weight-based caloric needs. The goal is to have 5 servings of vegetables, 2 fruits per day, and 5 vegetable color groups per week. Vegetables with high insoluble fiber content will be cooked instead of eaten raw.
  Interventions: Other: Anti-inflammatory diet
- Regular Diet (Active Comparator): Patients in the control diet arm will be counseled to continue their regular diets and focus on recording all food intake.
  Interventions: Other: Regular diet

INTERVENTIONS:
Other: Anti-inflammatory diet — Anti-inflammatory diet with increased vegetables, fruit, plant polyphenols, lean proteins, foods rich in omega-3s and unsaturated fats as well as decreased in processed refined foods.
  Arms: Anti-inflammatory whole food
Other: Regular diet — Focus on food journal and recording all food intake.
  Arms: Regular Diet

SUMMARY:
Patients with inflammatory bowel disease (IBD) often have narrowed microbial diversity and altered composition and function of the gut microbiome. We anticipate the anti-inflammatory diet, when compared with the usual diet, to produce favorable changes in these multi-omics profiles. These findings will provide insight into the interactions between diet and host biology, while providing clues on the mechanisms of diet therapy's effect and CD pathogenesis.

DETAILED DESCRIPTION:
A randomized controlled trial of the anti-inflammatory whole food diet versus usual diet for the induction of remission in 104 adults with mild-to-moderate Crohn's Disease (CD). The anti-inflammatory whole food diet will be compared to participants usual diet for understanding its effects on achieving clinical remission, clinical response, reduction in serological and fecal markers of inflammation, and improvement in patient-reported outcomes, such as physical activity, anxiety, depression, fatigue, pain, sleep disturbance, social satisfaction, and quality of life. The study will involve collection of blood and fecal specimens to evaluate the effects of the anti-inflammatory diet on the gut microbiome, bacterial metabolome, innate immune markers, and fecal microRNA profiles. The participants will be placed on anti-inflammatory diet for 8 weeks and assessed every 2 weeks for adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 75 years old
* History of Crohn's Disease (CD) with mild to moderate symptoms and prior biopsy proof

Exclusion Criteria:

1. History or current diagnosis of any of the following:

   * Stroke or Arrhythmia
   * Seizures
   * Liver Disease
   * Untreated hypertension (High Blood Pressure)
   * Active malignancy
   * Bleeding disorders
   * Heart Disease
   * Lung disease
   * Previous Heart surgery
   * Previous Gastrointestinal Surgery
   * Kidney Disease
   * Chronic Diarrhea
   * End enterostomy
   * Bulimia
   * Anorexia
   * Laxative Abuse
   * Endocrine Disorder
   * Current history of smoking tobacco
   * Urgent need for abdominal sugery
   * Severe Malnutrition
   * Active alcohol or non-cannabinoid substance abuse
2. Recent hospitalization within the last 30 days
3. Currently pregnant of lactating.
4. Current use probiotics or dietary supplements that would not be willing to discontinue for the length of the study.
5. Concerns for non-compliance
6. If currently on immunosuppressants, immunomodulators, cotticosteroids, and/or 5-aminosalicylates, no changes in doses will be permitted during the trial except for tapering of corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of the anti-inflammatory whole food diet for the induction of remission in Crohn's Disease | 8 weeks
  The patients' clinical response, defined by the Harvey-Bradshaw Index (HBI) (5 through 16 points) for clinical symptom improvement and/or remission.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Limketkai BN, Yang J, Chau L, Noorian S, Li Z. Randomized controlled trial of a natural whole food diet versus habitual diet for Crohn's disease: Is diet quality the key? Clin Nutr ESPEN. 2025 Oct;69:580-589. doi: 10.1016/j.clnesp.2025.08.015. Epub 2025 Aug 14. PMID 40818622